CLINICAL TRIAL: NCT06682845
Title: Association Between Drug-related Cutaneous Adverse Events and Progression Free Survival in Patients Treated with Enfortumab Vedotin
Acronym: SURVSKINTOX-EV
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0588
Record Dates: First submitted 2024-06-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Adverse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EV patients: Adult patients who have received enfortumab vedotin treatment at the Centre Léon Bérard or Hôpital Lyon Sud, and who do not object to the collection of their data.
  Interventions: Other: Collection of data in patients' medical files

INTERVENTIONS:
Other: Collection of data in patients' medical files — * Demographic data
  * Health data: body mass index, weight, tobacco consumption, history of hyperglycemia/ diabetes mellitus, Eastern Cooperative Oncology Group (ECOG) status, glomerular filtration rate, hemoglobin rate
  * Cancer-related data: date of diagnosis, tumoral site, tumor histology type, histology grade, date of first metastases involvement, presence of visceral metastases, presence of liver metastases, presence of lymph node-only metastases
  * Treatment-related data: previous line of treatment, co-treatment with anti-PD1, enfortumab vedotin (EV) treatment start date, EV treatment end date, EV posology, presence of EV reduction of dose or increased interval between perfusions, number of EV cycles
  * Adverse events (AE)-related data: occurrence of cutaneous AE, grade of cutaneous AE, date of cutaneous AE, type of cutaneous AE, management of cutaneous AE, discontinuation of EV treatment, rechallenge of EV treatment
  * Outcomes data: best overall response rate

SUMMARY:
Enfortumab vedotin (EV) is an antibody-drug conjugate (ADC) targeting nectin-4. In patients with metastatic urothelial carcinoma, EV in combination with pembrolizumab (anti-PD1) provides significantly better progression-free and global survival than platinum-based chemotherapies, with the benefit observed from the first line of treatment. However, EV is associated with a high frequency of cutaneous adverse events (AE), which may be due to physiological Nectin-4 expression in keratinocytes. These cutaneous toxicities include bullous/blistering toxicities and toxic epidermal necrolysis-like AE. While the association between cutaneous AE and survival has been demonstrated with anti-PD1, its association with survival in patient treated with ADC remains unknown. The objective of this retrospective dual-centric study is to determine whether there is an association between drug-related cutaneous AE and progression free survival in patients treated with EV.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients who have been treated with enfortumab vedotin at Hôpital Lyon Sud or Centre Léon Bérard and for whom follow-up data of at least 6 months are available are eligible for inclusion. To be included, patients must be willing and able to provide non-opposition consent for participation in this study and for the use of their medical data in this context.

Exclusion Criteria:

-Any medical, social, or psychiatric condition that might impair the patient's capacity to provide informed consent to participate in the study and to the use of their medical data is considered an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have received enfortumab vedotin treatment at the Centre Léon Bérard or Hôpital Lyon Sud, and who do not object to the collection of their data.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) according to the occurrence of cutaneous adverse events (AE) | From the start of EV treatment until disease progression or death, with data collected from 01/01/2015 to 02/05/2024.
  Progression-Free Survival (PFS) is defined as the time from the start of EV treatment to the occurrence of disease progression or death from any cause, whichever occurs first. This measure will assess the impact of any grade cutaneous adverse events (AEs) on PFS.

SECONDARY OUTCOMES:
Overall Survival (OS) according to the occurrence of cutaneous adverse events (AE) | From the start of EV treatment until death from any cause, with data collected from 01/01/2015 to 02/05/2024.
  Overall Survival (OS) is defined as the time from the start of EV treatment to death from any cause. This measure will assess the impact of any grade cutaneous adverse events (AEs) on OS.
PFS/OS according to blistering toxicity | From the start of EV treatment until disease progression, death, or first occurrence of blistering toxicity, with data collected from 01/01/2015 to 02/05/2024.
  This measure will assess PFS and OS in relation to the occurrence of blistering toxicity. Blistering toxicity is defined as a dermatosis with vesicular, bullous, and/or exfoliative lesions.
PFS/OS according to cutaneous AE in patients co-treated with anti-PD1 | From the start of combined EV and anti-PD1 treatment until disease progression or death, with data collected from 01/01/2015 to 02/05/2024.
  This measure will assess PFS and OS in relation to the occurrence of cutaneous adverse events in patients who are also receiving anti-PD1 treatment.
Identification of predictive risk factors for cutaneous AE | Retrospective analysis of data from the treatment initiation until the last recorded follow-up, with data collected from 01/01/2015 to 02/05/2024.
  Identification of potential predictive risk factors associated with the occurrence of cutaneous adverse events (defined as any grade skin rash, excluding isolated pruritus).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, Hospices Civils de Lyon, Oullins, France

IPD SHARING:
Plan to Share IPD: No